CLINICAL TRIAL: NCT00721851
Title: Coronary Artery Imaging With 320-slice Computed Tomography
Brief Title: 320-slice Coronary Computed Tomography (CT) Angiography
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Marc Dewey, Charité
Other Study IDs: EA1/140/07
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this study is to determine the potential utility of 320-slice volume-CT for obtaining adequate diagnostic accuracy while at the same time improving image quality compared with previous generations of CT scanners and simultaneously enabling a reduction in both radiation exposure and contrast agent amount required.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age
* sinus rhythm

Exclusion Criteria:

* prior conventional coronary angiography
* unstable presentation
* coronary artery bypass graft or stent
* pregnancy or breast-feeding
* creatinine > 2.0 mg per deciliter

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible patients referred to the Charité and scheduled to undergo conventional coronary angiography.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, MD, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Dewey M, Zimmermann E, Laule M, Rutsch W, Hamm B. Three-vessel coronary artery disease examined with 320-slice computed tomography coronary angiography. Eur Heart J. 2008 Jul;29(13):1669. doi: 10.1093/eurheartj/ehm626. Epub 2008 Feb 7. No abstract available. PMID 18263576
- [Background] Zimmermann E, Dewey M. Whole-heart 320-row computed tomography: reduction of radiation dose via prior coronary calcium scanning. Rofo. 2011 Jan;183(1):54-9. doi: 10.1055/s-0029-1245629. Epub 2010 Aug 19. PMID 20725881
- [Background] Dewey M, de Vries H, de Vries L, Haas D, Leidecker C. The present and future of cardiac CT in research and clinical practice: moderated discussion and scientific debate with representatives from the four main vendors. Rofo. 2010 Apr;182(4):313-21. doi: 10.1055/s-0029-1245195. Epub 2010 Mar 16. PMID 20234975
- [Result] Dewey M, Zimmermann E, Deissenrieder F, Laule M, Dubel HP, Schlattmann P, Knebel F, Rutsch W, Hamm B. Noninvasive coronary angiography by 320-row computed tomography with lower radiation exposure and maintained diagnostic accuracy: comparison of results with cardiac catheterization in a head-to-head pilot investigation. Circulation. 2009 Sep 8;120(10):867-75. doi: 10.1161/CIRCULATIONAHA.109.859280. Epub 2009 Aug 24. PMID 19704093